CLINICAL TRIAL: NCT02533856
Title: Randomized Control Trial of Emergency Department Discharge With Enhanced Transitions of Care Compared to Usual Care
Brief Title: Trial of Emergency Department Discharge With Enhanced Transitions of Care Compared to Usual Care
Acronym: ETOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15G.242
Record Dates: First submitted 2015-08-21; First posted 2015-08-27 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Patient Discharge; Emergency Care
MeSH Terms: interventions — d,d-T80-prallethrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Discharge from emergency department by usual care
- ETOC (Experimental): Discharge from emergency department with increased support services provided by BoardRounds after ED discharge
  Interventions: Other: ETOC

INTERVENTIONS:
Other: ETOC — Services provided to assist patients in accessing needed healthcare services after emergency department discharge such as scheduling appointments, finding new doctors, getting medications, or addressing problems with insurance coverage.
  Arms: ETOC

SUMMARY:
This is a randomized controlled trial to assess the relative effectiveness of providing Enhanced Transitions of Care (ETOC) to improve patient outcomes after discharge from the Emergency Department (ED). Patients who are being discharged from the ED and have had a previous ED visit or hospital admission within the Thomas Jefferson Hospital System (TJUH or Methodist) within the past 90 days will be eligible for enrollment in this trial. Patients who consent to enrollment will be randomized to discharge by usual care or discharge with ETOC as provided by the company BoardRounds.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 yrs and older) patients
* Have had a previous ED visit or hospital admission in the 90 days prior to the current ED visit (at Thomas Jefferson University Hospital or Methodist Hospital)
* Have just completed evaluation in the Thomas Jefferson University Hospital Emergency Department for any problem,
* Are ready for discharge from the Thomas Jefferson University Hospital ED, and
* Provide informed consent

Exclusion Criteria:

* Non-English speaking patients
* Patients undergoing medical clearance for a detox center or any involuntary court or magistrate order
* Patients who live outside Philadelphia area (unable to seek follow-up care in Philadelphia) or other condition known to preclude follow-up (such as no reliable access to a telephone)
* Patients in police custody or currently incarcerated individuals
* Patients who have, in their clinician's best judgment, major communication barriers such as visual or hearing impairment or dementia that would compromise their ability to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Total number of ED visits, hospital admissions, and outpatient office visits as determined by medical record review and patient report | 30 days
  30-day healthcare utilization will be measured by assessing the total number of ED treat-and-release visits, hospital admissions, and outpatient care visits in the 30 days after study enrollment - will be reported in aggregate and separately for each type of utilization (ED, inpatient hospital stay, office visit). Counts will be determined by medical record review for visits occurring within the health system, and will be supplemented by patient report in a 30-day survey to determine utilization outside the health system.

SECONDARY OUTCOMES:
Total number of ED visits, hospital admissions, and outpatient office visits as determined by medical record review and patient report | 9 days
  9-day healthcare utilization will be measured by assessing the total number of ED treat-and-release visits, hospital admissions, and outpatient care visits in the 30 days after study enrollment - will be reported in aggregate and separately for each type of utilization (ED, inpatient hospital stay, office visit). Counts will be determined by medical record review for visits occurring within the health system, and will be supplemented by patient report in a 30-day survey to determine utilization outside the health system.
Description of types of and count (per type) of assistance received by patients in accessing needed healthcare services as assessed by patient survey | 30 days
  Patients will be surveyed at 30 days to determine the types of assistance received, and frequency with which each type was received, in accessing needed healthcare services since their discharge from the ED.
Description of types of and count (per type) of assistance received by patients in accessing needed healthcare services as assessed by patient survey | 9 days
  Patients will be surveyed at 30 days to determine the types of assistance received, and frequency with which each type was received, in accessing needed healthcare services since their discharge from the ED.
Assessment of whether patient had unmet needs in accessing needed healthcare services, as determined by patient survey | 30 days
  Determination of whether patient had unmet needs (yes/no) in accessing needed healthcare services in the 30-days after ED discharge as identified by patient in a survey administered at 30 days post-discharge.
Assessment of whether patient had unmet needs in accessing needed healthcare services, as determined by patient survey | 9 days
  Determination of whether patient had unmet needs (yes/no) in accessing needed healthcare services in the 9-days after ED discharge as identified by patient in a survey administered at 9 days post-discharge.

OTHER OUTCOMES:
Description of unmet needs in accessing needed healthcare services as assessed in a patient survey | 30 days
  This will be a descriptive outcome to describe the types and counts of unmet needs that are identified by patients in the 30-days after ED discharge, as assessed in a survey administered 30 days after discharge. There will not be statistical analysis performed on this outcome, rather it will be descriptive and exploratory regarding patient primary struggles after ED discharge.